CLINICAL TRIAL: NCT06514612
Title: A Randomised, Double-Masked, Placebo-Controlled Phase 3 Study on the Efficacy and Safety of STN1013800 (Oxymetazoline HCl 0.1% Eye Drops) Used Twice Daily (BID) in the Treatment of Acquired Blepharoptosis
Brief Title: LIDRISE Study: A Phase 3 Study on the Efficacy and Safety of STN1013800 (Oxymetazoline HCl 0.1% Eye Drops, Single Dose) in the Treatment of Acquired Blepharoptosis.
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Santen SAS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 101380003SA
Record Dates: First submitted 2024-07-03; First posted 2024-07-23 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Acquired Blepharophimosis
MeSH Terms: interventions — Oxymetazoline; Ophthalmic Solutions

STUDY DESIGN:
Intervention Model Description: Subjects diagnosed with acquired blepharoptosis who meet eligibility criteria at Visit 1 (Screening) will return within 8 days for Visit 2 (Baseline, Day 1). At Visit 2 (Baseline, Day 1) they will be randomised to receive double-masked treatment for 6 weeks, with study visits completed at Week 2 (Day 14) and Week 6 (Day 42), and a post-treatment visit completed 2 weeks (± 3 days) after last study drug administration. This study will consist of a screening period of up to 8 days, a 6-week double-masked treatment period, and a post-treatment visit 2 weeks after the last administration of the study drug.
Who Masked: Participant, Care Provider, Investigator
Masking Description: This is a double -masked study with subjects, Investigators, Site Staff, Reading Centre personnel, and Santen personnel involved in the conduct of the study all masked to the study treatment.
  Each eligible subject will receive a numbered study treatment kit assigned by central randomisation via IWRS at Baseline.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- STN1013800 (0.1% Oxymetazoline Hydrochloride) eye drops in single dose containers (Experimental)
  Interventions: Drug: STN1013800 (0.1% Oxymetazoline Hydrochloride) eye drops in single dose containers
- Placebo (0% Oxymetazoline Hydrochloride) eye drops in single dose containers (Placebo Comparator)
  Interventions: Other: Placebo (0% Oxymetazoline Hydrochloride) eye drops in single dose containers

INTERVENTIONS:
Drug: STN1013800 (0.1% Oxymetazoline Hydrochloride) eye drops in single dose containers — STN1013800 (0.1% Oxymetazoline Hydrochloride) eye drops in single dose containers
  Arms: STN1013800 (0.1% Oxymetazoline Hydrochloride) eye drops in single dose containers
Other: Placebo (0% Oxymetazoline Hydrochloride) eye drops in single dose containers — Placebo (0% Oxymetazoline Hydrochloride) eye drops in single dose containers
  Arms: Placebo (0% Oxymetazoline Hydrochloride) eye drops in single dose containers

SUMMARY:
A Randomised, Double-Masked, Placebo-Controlled Phase 3 Study on the Efficacy and Safety of STN1013800 (Oxymetazoline HCl 0.1% Eye Drops) used twice daily (BID) in the Treatment of Acquired Blepharoptosis

DETAILED DESCRIPTION:
This is a randomised, double-masked, placebo-controlled Phase 3 study of the safety and efficacy of STN1013800 in the treatment of acquired blepharoptosis.

Subjects diagnosed with acquired blepharoptosis who meet eligibility criteria at Visit 1 (Screening) will return within 8 days for Visit 2 (Baseline, Day 1). At Visit 2 (Baseline, Day 1) they will be randomised to receive double-masked treatment for 6 weeks, with study visits completed at Week 2 (Day 14) and Week 6 (Day 42), and a post-treatment visit completed 2 weeks (± 3 days) after last study drug administration. Approximately 234 adult subjects with blepharoptosis who meet all the eligibility criteria will be randomised in a 1:1 ratio to receive:

* STN1013800 BID
* Placebo BID

Note that:

* On study visits Day 1 and Day 42, the AM dose is administered at 08:00 (at site) and the PM dose is administered at 16:00 (self-administered at home)
* On study visit Day 14, the AM dose is administered at 06:00 (self-administered at home), the PM dose is administered at 14:00 (at site)

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and sign an informed consent form prior to participation in any studyrelated procedures.
* Male or female subjects ≥ 18 years and ≤ 75 years.
* Presence of all the following at Screening:

  1. diagnosis of acquired ptosis in both eyes with MRD 1 ≥0 and ≤ 2 mm in the study eye
  2. Snellen VA of 20/80 or better in both eyes Note: MRD1 is defined as the distance between upper eye lid margin and centre of the pupil. MRD0 is defined as the upper eye lid margin at the centre of the pupil. Measurement of MRD1 will be done by a Central Reading Centre. If the centre of the pupil cannot be determined by the Central Reading Centre due to negative MRD1, the subject will be deemed ineligible.
* Females who are 1-year postmenopausal, surgically sterilised, or females of childbearing potential with a negative urine pregnancy test at screening (Visit 1). Females of childbearing potential must use an acceptable form of contraception throughout the study. Acceptable methods include the use of at least one of the following: intrauterine (intrauterine device), hormonal (oral, injection, patch, implant, ring), barrier with spermicide (condom, diaphragm), or abstinence.
* A male subject with a female partner of childbearing potential should use or practice an acceptable contraceptive method, such as abstinence, condom or vasectomy (surgery at least 6 months prior to signing the study ICF and beginning screening), or other contraception deemed adequate by the investigator during the study.
* Able to self-administer study treatment or to have the study treatment administered by a caregiver throughout the study period.
* An answer of 'Yes' to the question 'Does the ptosis cause enough burden to the subject to want to receive treatment for it'.
* Loss of ≥ 8 points not seen at or above 10° from fixation in the superior visual field of a reliable HVF 36-point ptosis protocol test at screening visit in the same eye with MRD1 ≥0 and ≤ 2 mm. If both eyes have MRD1 ≥0 and ≤ 2 mm the more ptotic eye (the eye with the smaller MRD1 measurement) will be the study eye. If the MRD1 is the same in both eyes, the eye with the worse VF will be the study eye. If the MRD1 and VF is the same in both eyes, the right eye will be the study eye. The HVF Analyzer will determine if the visual field test is reliable. If the HVF Analyzer issues an "XX" for fixation losses, false positives, and/or false negatives, the test will be deemed unreliable. If deemed unreliable, the test must be retaken once per scheduled screening visit. If a reliable visual field cannot be obtained, the subject will be a screen failure.

Exclusion Criteria:

* In either eye:
* Congenital ptosis.
* Presence of either of the following:

  1. Pseudo ptosis (upper eyelid dermatochalasis that overhangs the upper eyelid margin); or
  2. Dermatochalasis that extends less than 3 mm above the upper eyelid margin.
* Neurogenic ptosis (e.g., Horner's syndrome, 3rd cranial nerve palsy).
* Myogenic ptosis.
* Marcus Gunn jaw-winking syndrome.
* Previous ptosis surgery (previous blepharoplasty is allowed provided the surgery took place at least 3 months prior to screening [Visit 1]).
* Lid position affected by lid or conjunctival scarring.
* Visual field loss from any cause other than ptosis.
* History of herpes keratitis.
* Poor fixation or abnormal eye position which prevents from taking reliable pictures for MRD1 measurement.
* History of closed/narrow angle glaucoma (unless patent peripheral iridotomy has been performed at least 3 months prior to screening (Visit 1).
* Facial including periocular neurotoxin (e.g., Botox, Xeomin, Dysport, Myobloc) injections within 3 months prior to screening (Visit 1) and during the study.
* Topical application of bimatoprost (i.e., Latisse®) to the eyelashes within 8 days prior to screening (Visit 1) and during the study.
* Mechanical ptosis e.g., ptosis due to orbital, corneal or lid tumor, cicatricial processes affecting the movements of the upper lid, and enophthalmos.
* Use of topical ophthalmic medications including anti-allergy [e.g., antihistamines], dry eye medications [e.g., IKERVIS®] (except artificial tears with anticipated stable usage during the study), antimicrobial drugs [e.g., antibiotics and antivirals], and anti-inflammatory drugs [including nonsteroidal anti-inflammatory drugs (NSAIDs) and steroids] within 8 days prior to screening (Visit 1) and during the study. Timolol maleate, or sympathetic alpha receptor agonists (e.g., brimonidine tartrate, or apraclonidine hydrochloride) for the treatment of elevated intraocular pressure. Please note that topical ophthalmic prostaglandin analogues for the treatment of elevated intraocular pressure are permitted if dosed in the evening in accordance with the approved prescribing information. All other topical antiglaucoma medications are prohibited.
* Any intravitreal injections (e.g., antiVEGFs, steroids) within 8 days prior to screening (Visit

  1) and during the study.
* Current punctal plugs or placement of punctal plugs during the study.
* Current use of OTC vasoconstrictor/decongestant eye medication (e.g., Visine® L.R.®) or any ophthalmic or non-ophthalmic α-adrenergic agonist including OTC products (e.g., Afrin®) at any time during the study, (artificial tears are allowed).
* Monoamine oxidase inhibitors (MAOI) (e.g., selegiline hydrochloride, rasagiline mesilate, safinamide mesilate).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Estimated)
Dates: Start 2024-12-30 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Marginal Reflex Distance (MRD1) on Day 14 at 4 hours after PM dose. | Day 14 at 4 hours
  Change from baseline in MRD1 (Marginal Reflex Distance, Distance from the centre of the pupil to central upper lid margin) on Day 14 at 4 hours after PM dose. This is to evaluate the efficacy of STN1013800 dosed twice daily in the treatment of acquired blepharoptosis on Day 14

SECONDARY OUTCOMES:
PRO (Patient Reported Outcome): PGIC (Subject Global Impression of Change) on Day 14, 4 hours after PM dose | Day 14 at 4 hours
  To assess the degree of improvement experienced by subjects since start of the trial (PRO)

CONTACTS AND LOCATIONS:
Locations (37):
- Czechia (3):
  - Oftex.s.r.o, oční klinika, Pardubice
  - Fakultni nemocnice Plzeň, Oční oddělení, Pilsen
  - Fakultni Thomayerova nemocnice, Prague
- France (4):
  - Clinique Ophtalmologique Thiers, Bordeaux
  - CHU Rennes - PONTCHAILLOU Service ophtalmologie, Guillon
  - Hôpital Fondation Adolphe de Rothschild, Paris
  - CHU de Saint Etienne - Hôpital NORD Service d'Ophtalmologie, Saint-Etienne
- Germany (2):
  - Unversitaetsmedizin Goettingen, Goettigen
  - Universitätsmedizin Göttingen; Georg-August-Universität, Göttingen
- Hungary (5):
  - Budapest Retina Associates, Budapest
  - Budapesti Jahn Ferenc Dél-Pesti Kórház és Rendelőintézet, Budapest
  - Észak-Pesti Centrumkórház - Honvédkórház, Budapest
  - Debreceni Egyetem Klinikai Központ, Debrecen
  - Ganglion Orvosi Központ - Nozologen Kft., Pécs
- Italy (3):
  - AOU di Ferrara, Arcispedale Sant'Anna, Ferrara
  - AOU Federico II, Napoli
  - PU A. Gemelli, Università Cattolica del Sacro Cuore, Roma
- Netherlands (2):
  - Leiden University Center (LUMC), Leiden
  - Oogziekenhuis Rotterdam, Rotterdam
- Poland (5):
  - Profesorskie Centrum Okulistyki OKULISTYKA OPTIMUM, Gdansk
  - Gabinet Okulistyczny Prof. Edward Wylegala, Katowice
  - Centralny Szpital Kliniczny MSWiA w Warszawie, Oddzial Okulistyki, Warsaw
  - Military Institute of Medecine - National Institute of Research, Oddzial Okulistyki, Warsaw
  - Military Institute of Medecine - National Institute of Research, Warsaw
- Spain (7):
  - Hospital Universitario Virgen de las Nieves, Granada
  - Virgen de las Nieves University Hospital, Granada
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario Ramón y Caja, Madrid
  - Complexo Hospitalario Universitario de Santiago, Santiago de Compostela
  - Hospital Universitario Miguel Servet, Zaragoza
  - Miguel Servet University Hospital, Zaragoza
- United Kingdom (6):
  - Leeds Teaching Hospitals NHS Trust, St James's University Hospital, Leeds
  - Moorfields Eye Hospital NHS Foundation Trust - Moorfields Eye Hospital, London
  - FaceRestoration Ltd, London
  - Opal Clinic London Ltd, London
  - South tyneside & Sunderland NHS Trust, Sunderland Eye Infirmary, Sunderland
  - South Tyneside and Sunderland NHS Foundation Trust, Sunderland Eye Infirmary, Sunderland